CLINICAL TRIAL: NCT02450487
Title: Influence of Genotype of Cytochrome P450 (CYP2C9) on Clinical Efficacy and Pharmacokinetics of Piroxicam After Lower Third Molar Surgery
Brief Title: Influence of Genotype of CYP2C9 on Clinical Efficacy and Pharmacokinetics of Piroxicam After Lower Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Adriana Maria Calvo, PhD DDS, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20657913.7.0000.5417 CAAE
Record Dates: First submitted 2015-05-15; First posted 2015-05-21 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Pain; Other Surgical Procedures; Impacted Third Molar Tooth; Cytochrome P450 CYP2C9 Enzyme Deficiency
Keywords: Piroxicam; Pharmacogenetic; Lower Third molar
MeSH Terms: conditions — Pain | interventions — Piroxicam; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional group (Experimental): 100 patients will be treated with Piroxicam (20 mg once daily for 4 days) for pain control after lower third molar surgery
  Interventions: Drug: Piroxicam

INTERVENTIONS:
Drug: Piroxicam — After extraction of at least one third molar, 100 patients will be treated with Piroxicam (20 mg once daily for 4 days) for pain control, collect the saliva to be genotyped and phenotyped for CYP2C9 (by PCR) and their post-operative notes (pain, swelling, trismus, temperature) will be analyzed. For the pharmacokinetics of piroxicam saliva samples will be collected from 10 of these patients at different times after ingestion of a capsule of 20 mg Piroxicam (before, 1, 2, 3, 4, 5, 6, 8, 11, 24, 48 and 72 hours after ingestion).
  Other Names: Lower third molar surgery; Pharmacogenetics

SUMMARY:
Pharmacogenetics is an area of Pharmacology that studies the contribution of genetic factors to individual responses to drugs. This branch of science involves the variability in pharmacodynamics and pharmacokinetics through the study of polymorphisms in genes encoding receptors, as well as in drug metabolism, where this area of Pharmacology has been growing and achieving its first results with clinical use. The non-steroidal anti-inflammatory (NSAIDS) are metabolized by cytochrome P450 (CYP) family, predominantly CYP2C9. The goal of this study is to evaluate the different gene haplotypes for the clinical efficacy of piroxicam after third lower molar surgery for pain, edema and trismus, adverse reactions, need of rescue medication, patient satisfaction regarding the drug and the pharmacokinetics of the drug between the different gene haplotypes for CYP2C9 that are found in this population. Therefore, 60 patients will be genotyped and phenotyped for this gene and their postoperative data will be confronted with the data found in the Brazilian population. For the analysis of the proposed gene, saliva will be collected and serve as a source of genomic DNA. For the molecular analysis, polymerase chain reaction (PCR) with tests validated and produced by Applied Biosystems® will be performed. For the pharmacokinetics, saliva samples will be collected at various times according to protocols available in the literature, and piroxicam concentrations in the samples will be measured by high pressure liquid chromatography (HPLC) and Liquid chromatography-mass spectrometry (LC MS/MS). The analysis of the results will be described with a significance level of 0.05.

DETAILED DESCRIPTION:
Lower third molars (with high degree of difficulty) surgeries will be performed in Clinical Pharmacology Laboratory at the Bauru School of Dentistry - University of São Paulo (FOB-USP), which will be provided to patients daily doses of piroxicam 20 mg 4 days. Thus collect data related to pain, swelling, trismus, amount of rescue medication required by patients, overall assessment and satisfaction about taking medicine, saliva samples for the analysis of the pharmacokinetics of the drug, genotyping and phenotyping of the subjects of the research.

The global clinical evaluation along with genotyping and phenotyping these individuals can show us if there is an influence not only in adverse effects, but also in the therapeutic effects of the drug in the Brazilian population. Research of this nature are rare in this area of Clinical Pharmacogenetics and can be of great help in prescribing these drugs to control pain and inflammation.After the removal of third molars will make collecting 6 mL of saliva in several post-surgical moments for analysis of the pharmacokinetics of the drug piroxicam and 10 mL of saliva for the analysis of genetic material. It is noteworthy that this project will initiate the nucleation of a new line of research in college, the first in Pharmacogenetics area conducted in FOB / USP.Will be assessed the following parameters in all patients after surgery of at least a third lower molar with a high degree of difficulty (Annexes 1, 2 and 3): 1) onset and duration of surgery after the administration of the local anesthetic, 2) open mouth prior to surgery, on the 2nd day after the surgery and on the 7th day after surgery (removal of stitches); 3) measured the facial edema in the second day after surgery and on the 7th day after surgery (compared to the measurements obtained before surgery); 4) body temperature before surgery, on the 2nd day after the operation and on the 7th day after surgery (removal of stitches); 5) incidence, type and severity of adverse reactions, 6) plug pain (VAS - visual analog scale) filled by patients for 4 days after prescription Piroxicam; 7) amount of rescue medication required by patients.

The comparative analysis of the data, along with data on the pharmacokinetics of the drug, genotyping and phenotyping the CYP2C9 gene, provide the basis for evaluation of the influence of the gene in clinical efficacy, side effects and need for relief medication required by patients after surgery third- molars with a high degree of difficulty, which was prescribed as anti-inflammatory piroxicam.

ELIGIBILITY:
Inclusion Criteria:

* Impacted lower third molar;
* not making use of nonsteroidal anti-inflammatory drugs in the last 7 days;

Exclusion Criteria:

* Local anesthetics allergy;
* History of gastrointestinal bleeding or ulcers;
* Kidney disease;
* Asthma;
* Allergy or sensitivity to aspirin or any other anti-inflammatory non-steroid agent;
* Pregnant or nursing women;
* Patients using antidepressant, diuretic or aspirin;
* Patients received antibiotics for 30 days prior to surgery.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Calvo, PhD, Study Chair — Bauru School of Dentistry/University of Sao Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventional Group: 102 patients were treated with Piroxicam (20 mg once daily for 4 days) for pain control after lower third molar surgery
  Piroxicam: After extraction of at least one third molar, 102 patients were treated with Piroxicam (20 mg once daily for 4 days) for pain control, collected saliva to be genotyped and phenotyped for CYP2C9 (by PCR) and their post-operative notes (pain, swelling, trismus, temperature) were analyzed. For the pharmacokinetics of piroxicam saliva samples were collected from 10 of these patients at different times after ingestion of a capsule of 20 mg Piroxicam (before, 1, 2, 3, 4, 5, 6, 8, 11, 24, 48 and 72 hours after ingestion).
Period: Overall Study
Arm/Group | Interventional Group
Started | 105
Completed | 102
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Interventional Group
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 102

OUTCOME MEASURES:

1. Primary Outcome: Score of Pain Measured by Visual Analogue Scale
Description: Score of pain after third molar surgery is measured by visual analogue scale (0-100mm).
Time Frame: at 24 hours after surgery
Population: Pain control was measure at 24h after surgery
Measure: Mean (Standard Deviation); unit: score on a scale (mm)
Groups:
- Interventional Group: After extraction of one lower third molar, 102 patients were treated with Piroxicam (20 mg once daily for 4 days) for pain control
Arm/Group | Interventional Group
Number analyzed (Participants) | 102
score on a scale (mm) | 25 (25)

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Report of adverse effects during the postoperative period until suture removal seven days after extraction of third molar included and/or impacted in patients underwent surgery.
Time Frame: Seven days after surgery
Population: Throughout the entire study, only two volunteers reported adverse side effects; on the second day, one volunteer reported sleepiness (CYP2C8*3 mt and CYP2C9*1/*3 genotype) and one volunteer (CYP2C8*3 mt and CYP2C9*1/*3 genotype) reported stomachaches.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Group
Number analyzed (Participants) | 102
Participants | 2

ADVERSE EVENTS:
Time Frame: 7 days post-operatively
Description: sleepiness and stomachaches.
Arm/Group | Interventional Group
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 2/102
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Group (N=102)
Sleepness (Nervous system disorders) | 1 (1) — on the second day, one volunteer reported sleepiness (CYP2C8*3 mt and CYP2C9*1/*3 genotype)
Stomachaches (Gastrointestinal disorders) | 1 (1) — one volunteer (CYP2C8*3 mt and CYP2C9*1/*3 genotype) reported stomachaches

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No